CLINICAL TRIAL: NCT01605539
Title: Cannabidiol as Treatment Intervention for Opioid Relapse
Brief Title: Acute and Short-term Effects of Cannabidiol Admin on Cue-induced Craving in Drug-abstinent Heroin Dependent Humans
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hurd,Yasmin, Ph.D. (Individual)
Responsible Party: Principal Investigator, Yasmin Hurd, Principal Investigator, Hurd,Yasmin, Ph.D.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R21 DA027781(2); R21DA027781 (NIH)
Record Dates: First submitted 2012-05-02; First posted 2012-05-25 (Estimated); Results first posted 2016-11-28 (Estimated); Last update posted 2020-08-11 (Actual); Status verified 2020-07

CONDITIONS: Opiate Addiction
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Placebo Comparator): Subjects will receive pills that resemble the Cannabidiol capsule but do not have have its properties.
  Interventions: Drug: Control
- Cannabidiol 400 (Experimental): Subjects in Arm Cannabidiol 400 will receive 400 mg of cannabidiol
  Interventions: Drug: Cannabidiol 400
- Cannabidiol 800 (Experimental): Subjects in Arm Cannabidiol 800 will receive 800mg of cannabidiol
  Interventions: Drug: Cannabidiol 800

INTERVENTIONS:
Drug: Cannabidiol 400 — Subjects in Arm CBD 400 will receive 400mg of Cannabidiol in each of the three test sessions
  Other Names: CBD
  Arms: Cannabidiol 400
Drug: Cannabidiol 800 — Subjects in Arm CBD 800 will receive 800mg of Cannabidiol in each of the three test sessions
  Other Names: CBD
  Arms: Cannabidiol 800
Drug: Control — Subjects will receive a harmless, inactive pill to compare and validate the results of the other arms of the study
  Other Names: CBD
  Arms: Control

SUMMARY:
Despite the current available therapies for opioid-dependent patients, most patients relapse. This research project focuses on the development of a novel compound, cannabidiol, to modulate opioid craving in humans based on animal models showing its selective effectiveness to inhibit drug-seeking behavior. The development of a targeted treatment for opioid relapse would be of tremendous medical and public health value.

DETAILED DESCRIPTION:
Opioid abuse is a significant global public health problem. Of the more than one million people suffering today from opiate dependency, less than a quarter of such individuals receive treatment. Pharmacotherapeutic approaches traditionally have targeted mu opioid receptors since heroin and its metabolites bind with highest affinity to this receptor subtype. Although such treatment strategies have improved substance abuse outcomes, they do not effectively block opiate craving and thus are still associated with high rates of relapse. Using a strategy of indirectly regulating neural systems to modulate opioid-related behavior, our preclinical rodent studies consistently demonstrated that cannabidiol (CBD), a nonpsychoactive component of cannabis, specifically inhibited cue-induced heroin-seeking behavior. CBD's selective effect on drug-seeking behavior was pronounced after 24 hrs and endured even two weeks after the last drug administration following short-term CBD exposure. The fact that drug craving is generally triggered by exposure to conditioned cues suggests that CBD might be an effective treatment for heroin craving, specially given its protracted impact on behavior. CBD has already been shown in Phase I of our study and in various clinical studies to be well tolerated with a wide safety margin in human subjects. CBD thus represents a strong candidate for the development as a potential therapeutic agent in humans for opioid craving and relapse prevention. It is the goal of this second exploratory phase of the project to characterize the effects of CBD administration on cue-induced craving in drug-abstinent heroin-dependent subjects using a random double blind design during a post-acute (greater than 6 days since last use) heroin withdrawal period. Study participants will be administered CBD during 3 test sessions and studied for the effects on cue-induced craving during those sessions as well as one week after the final CBD administration on the final test day (session 4).

ELIGIBILITY:
Inclusion Criteria:

* Must be between 21 and 65 years old
* Must have an opiate dependence that meets criteria set in the Structured Clinical Interview for DSM-IV(SCID-IV) over the last three months
* No opioid use in the past 7 days (will be verified via urine drug screen and opiate metabolite test)

Exclusion Criteria:

* Using any psychoactive drug (other than nicotine) any time up to test session 3
* Having a diagnosis of drug dependence (except for heroin or nicotine) in the past 3 months, based on the SCID-IV interview criteria
* Being maintained on methadone or buprenorphine, or taking opioid antagonists such as naltrexone
* Having a positive a drug screen
* Showing signs of acute heroin withdrawal symptoms
* Having medical conditions, including Axis I psychiatric conditions under DSM-IV (examined using the Mini International Neuropsychiatric Interview [MINI])
* Having a a history of cardiac disease, arrhythmias, head trauma, and seizures
* Having a history of hypersensitivity to cannabinoids
* Arriving to the study site visibly intoxicated as determined by a clinical evaluation for signs and symptoms of intoxication and as verified by a drug screen
* Participating in a another pharmacotherapeutic trial in the past 3 months
* Being pregnant of breastfeeding
* Not using or irregularly using appropriate methods of contraception such as hormonal contraceptives (e.g., Depo-Provera, Nuva-Ring), an intrauterine device (IUD), or double barrier method (combination of any two barrier methods used simultaneously, e.g., condoms, spermicide, diaphragms)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-05; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yasmin Hurd, Ph.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- CBD 400 Group: Subjects will receive 400 mg of cannabidiol
  Subjects in Arm CBD 400 will receive 400 mg of Cannabidiol in each of the three test sessions
- CBD 800 Group: Subjects in Arm CBD 800 will receive 800 mg of Cannabidiol in each of the three test sessions
Period: Overall Study
Arm/Group | Control | CBD 400 Group | CBD 800 Group
Started | 3 | 3 | 4
Completed | 3 | 2 | 4
Not Completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control: Subjects received pills that resemble the Cannabidiol capsule but did not have its properties.
  Control: Subjects receivd a harmless, inactive pill to compare and validate the results of the other arms of the study
- CBD Group: The two arms (400 mg and 800 mg of Cannabidiol) were combined for analysis because the sample size was too small and dividing the two arms would not have yielded a meaningful analysis.
  Cannabidiol: Subjects in Arm CBD Group received 400 mg or 800mg of Cannabidiol in each of the three test sessions
- Total: Total of all reporting groups
Arm/Group | Control | CBD Group | Total
Number analyzed (Participants) | 3 | 6 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 6 | 9
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 6 | 9
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Changes in Cue-Induced In-Clinic Craving (From Baseline to Post-cue or Post-neutral - Via the Visual Analog Scale for Craving (VASC)
Description: The VASC will be administered to assess potential variations in the subjective craving effects associated with heroin. Following the administration of the investigational drug, craving induced in response to the cue sessions and neutral cue sessions in the clinic will be measured. In this way, changes in craving from baseline (pre-cue to post-cue and pre-neutral cue to post-neutral cue) within each test visit) will be measured and compared. Scale range: 0 (no craving) - 10 (extreme craving).
  **For test visits I, II and IV, there will be two cue sessions at each test visit: a neutral cue video (PN) and a drug-related cue video (PC) will be shown in random order at each visit. Before the beginning of each cue session (PN or PC), baseline measures will be taken. The same questionnaires will be administered immediately following the neutral cue video and the drug-related cue video. Thus there will be two sets of baselines and two sets of post cue measurements per test visit for test
Time Frame: VASC: test visits I, II and IV - baseline 1, post cue (PC), baseline 2, post neutral cue (PN)
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Control: Subjects received pills that resemble the Cannabidiol capsule but do not have have its properties.
  Control: Subjects received a harmless, inactive pill to compare and validate the results of the other arms of the study
- CBD Group: Subjects received 400 mg or 800mg of cannabidiol.The two arms (400 mg and 800 mg CBD groups) were combined for analysis as CPD Group because the sample size was too small and dividing the two arms would not have yielded a meaningful analysis.
  Cannabidiol: Subjects in Arm CBD Group received 400 mg or 800mg of Cannabidiol in each of the three test sessions
Arm/Group | Control | CBD Group
Number analyzed (Participants) | 3 | 6
units on a scale
  Test 1: Baseline to Post Drug Cue | 2.67 (1.45) | 0.83 (0.31)
  Test 1: Baseline to Post Neutral Cue | -0.33 (0.33) | -0.17 (0.17)
  Test 2: Baseline to Post Drug Cue | 0.670 (0.33) | 0.67 (0.71)
  Test 2: Baseline to Post Neutral Cue | -0.33 (0.67) | -0.67 (0.71)
  Test 4: Baseline to Post Drug Cue | 0.33 (0.33) | 0.33 (0.21)
  Test 4: Baseline to Post Neutral Cue | 1.00 (0.58) | -0.50 (0.22)

2. Primary Outcome: Changes in Out-of-Clinic Craving (From Pre-Dose to Approximately 6 Hours Post-Dose for Test Visits I and II; and From Pre-Dose Test Visit I to Pre-Cue Test Visit IV) - Via the Heroin Craving Questionnaire (HCQ)
Description: Subjects will be asked to complete the short version of the HCQ on their own time at home and bring it with them when they return for their next visit. Upon arrival to the clinic, subjects will also complete an HCQ with the coordinator to assess daily baseline cravings. This questionnaire will help us assess changes in craving generated outside of the clinical laboratory session from test visit 1 through test visit 4. Scale: 1 (strongly disagree) - 7 (strongly agree). Total Score Range: 14 (less cravings) - 98 (more cravings).
  ** The baseline measure for this outcome will be measured at the beginning of test session I prior to the administration of CBD/Placebo. Test measures will be taken approximately 6 hours following each dose for test sessions I, II and III. The final measure will be taken at test session IV, at the beginning of the session.
Time Frame: Test I and II: Change from pre-dose to approx. 6 hours post-dose; Change from pre-dose test visit I to pre-cue test visit IV
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Control: Subjects received pills that resembled the Cannabidiol capsule but did not have have its properties.
  Control: Subjects received a harmless, inactive pill to compare and validate the results of the other arms of the study
- CBD Group: Subjects received 400 mg or 800mg of cannabidiol. The two arms (400 mg and 800 mg CBD groups) were combined for analysis as CPD Group because the sample size was too small and dividing the two arms would not have yielded a meaningful analysis.
  Subjects in Arm CBD will receive 400 mg or 800mg of Cannabidiol in each of the three test sessions
Arm/Group | Control | CBD Group
Number analyzed (Participants) | 3 | 6
units on a scale
  Test 1: Change from pre-dose to 6 hrs post-dose | -3.67 (2.73) | -0.33 (3.57)
  Test 2: Change from pre-dose to 6 hrs post-dose | -5.33 (15.43) | -6.17 (1.11)
  Change from Test 1 (pre-dose) to Test 4 (pre-cue) | -4.33 (7.69) | -16.33 (3.97)

3. Secondary Outcome: Vital Signs - Blood Pressure
Description: Blood pressure (mmHg) will be monitored throughout the time course of the study and changes from baseline will be studied across the various time points.
  **For test visits I, II and IV, there will be two cue sessions at each test visit: a neutral cue video (PN) and a drug-related cue video (PC) will be shown in random order at each visit. Before the beginning of each cue session (PN or PC), baseline measures will be taken. Blood pressure will be measured again following the neutral cue video and the drug-related cue video. Thus there will be two sets of baselines and two sets of post cue measurements per test visit for test visits I, II and IV.
Time Frame: Test sessions 1,2,and 4: baseline 1, post cue (PC), baseline 2, post neutral cue (PN)
Measure: Mean (Standard Error); unit: mmHg
Groups:
- CBD Group: Subjects received 400 mg or 800mg of cannabidiol. The two arms (400 mg and 800 mg CBD groups) were combined for analysis as CPD Group because the sample size was too small and dividing the two arms would not have yielded a meaningful analysis.
  Subjects in Arm CBD received 400 mg or 800mg of Cannabidiol in each of the three test sessions
Arm/Group | Control | CBD Group
Number analyzed (Participants) | 3 | 6
mmHg
  Systolic BP change (mmHG): test 1, baseline to PC | 8.33 (3.76) | 4.5 (3.66)
  Systolic BP change (mmHG): test 1, baseline to PN | -0.33 (1.20) | 0.17 (3.60)
  Systolic BP change (mmHG): Test 2, baseline to PC | -8.67 (5.17) | 8.5 (5.37)
  Systolic BP change (mmHG): test 2, baseline to PN | 5.00 (3.79) | 4.83 (3.78)
  Systolic BP change (mmHG): Test 4, baseline to PC | 1.00 (2.52) | -6.33 (4.65)
  Systolic BP change (mmHG): test 4, baseline to PN | -11.67 (4.06) | 9.67 (6.23)
  Diastolic BP change (mmHG): test 1, baseline to PC | 6.33 (1.33) | 5.33 (2.63)
  Diastolic BP change (mmHG): test 1 baseline to PN | -0.33 (2.19) | 1.5 (2.51)
  Diastolic BP change (mmHG): test 2 baseline to PC | -4 (2.65) | 1.83 (3.33)
  Diastolic BP change (mmHG): test 2 baseline to PN | 3.67 (3.93) | 0.83 (2.20)
  Diastolic BP change (mmHG): test 4 baseline to PC | -0.33 (1.45) | 0.67 (3.34)
  Diastolic BP change (mmHG): test 4 baseline to PN | -3.67 (4.91) | -1.33 (4.62)

4. Secondary Outcome: Visual Analog Scale for Anxiety (VASA)
Description: Questionnaires will be used to measure subjective responses. Anxiety will be assessed using a visual analog scale for anxiety (VASA). Scale: 0 (not at all anxious) - 10 (extremely anxious).
  **For test visits I, II and IV, there will be two cue sessions at each test visit: a neutral cue video (PN) and a drug-related cue video (PC) will be shown in random order at each visit. Before the beginning of each cue session (PN or PC), baseline measures will be taken for each variable. The same variables will be measured following the neutral cue video and the drug-related cue video. Thus there will be two sets of baselines and two sets of post cue measurements per test visit for test visits I, II and IV.
Time Frame: Test visit I, II and IV: baseline 1, post cue (PC), baseline 2, post neutral cue (PN)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Control | CBD Group
Number analyzed (Participants) | 3 | 6
units on a scale
  Test 1: Baseline to Post Drug Cue | 2.00 (1.15) | 0.00 (0.26)
  Test 1: Baseline to Post Neutral Cue | 0.33 (0.33) | -0.33 (0.21)
  Test 2: Baseline to Post Drug Cue | 1.33 (1.20) | -0.50 (0.34)
  Test 2: Baseline to Post Neutral Cue | -0.67 (0.88) | -0.50 (0.34)
  Test 4: Baseline to Post Drug Cue | 0.00 (0.00) | 0.00 (0.00)
  Test 4: Baseline to Post Neutral Cue | -0.67 (0.67) | -0.33 (0.21)

5. Secondary Outcome: The Positive and Negative Affect Schedule (PANAS) - Positive Affect Schedule (PAS) Data
Description: Questionnaires will be used to measure subjective responses. The Positive and Negative Affect Schedule will allow us to obtain positive and negative affect measures and observe their changes from baseline over the course of the cue-induced craving session. Scale: 0 (only slightly or not at all) - 5 (extremely). Total Score Range for Positive Affect Assessment (PAS): 10 (minimum) - 50 (maximum). Higher score reflects stronger positive affect.
  **For test visits I, II and IV, there will be two cue sessions at each test visit: a neutral cue video (PN) and a drug-related cue video (PC) will be shown in random order at each visit. Before the beginning of each cue session (PN or PC), baseline measures will be taken for each variable. The same variables will be measured following the neutral cue video and the drug-related cue video. Thus there will be two sets of baselines and two sets of post cue measurements per test visit for test visits I, II and IV.
Time Frame: Test session 1, 2, and 4: baseline 1, post cue (PC), baseline 2, post neutral cue (PN)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Control | CBD Group
Number analyzed (Participants) | 3 | 6
units on a scale
  Test 1: Baseline to Post Drug Cue | 1.33 (2.40) | -0.50 (1.88)
  Test 1: Baseline to Post-Neutral Cue | 1.33 (1.20) | -1.83 (0.83)
  Test 2: Baseline to Post Drug Cue | -4.00 (1.73) | -1.00 (1.03)
  Test 2: Baseline to Post Neutral Cue | -4.67 (2.40) | 0.17 (1.01)
  Test 4: Baseline to Post Drug Cue | -3.50 (3.50) | -1.33 (0.61)
  Test 4: Baseline to Post Neutral Cue | 2.50 (2.50) | 0.67 (0.49)

6. Secondary Outcome: The Positive and Negative Affect Schedule (PANAS) - Negative Affect Schedule (NAS) Data
Description: Questionnaires will be used to measure subjective responses. The Positive and Negative Affect Schedule will allow us to obtain positive and negative affect measures and observe their changes from baseline over the course of the cue-induced craving session. Scale: 0 (only slightly or not at all) - 5 (extremely). Total Score Range for Negative Affect Assessment (NAS): 10 (minimum) - 50 (maximum). Higher score reflects stronger negative affect.
  **For test visits I, II and IV, there will be two cue sessions at each test visit: a neutral cue video (PN) and a drug-related cue video (PC) will be shown in random order at each visit. Before the beginning of each cue session (PN or PC), baseline measures will be taken for each variable. The same variables will be measured following the neutral cue video and the drug-related cue video. Thus there will be two sets of baselines and two sets of post cue measurements per test visit for test visits I, II and IV.
Time Frame: Test session 1, 2, and 4: baseline 1, post cue (PC), baseline 2, post neutral cue (PN)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Control | CBD Group
Number analyzed (Participants) | 3 | 6
units on a scale
  Test 1: Baseline to Post Drug Cue | 4.00 (3.51) | 0.50 (0.92)
  Test 1: Baseline to Post Neutral Cue | 1.33 (0.88) | -1.50 (0.67)
  Test 2: Baseline to Post Drug Cue | 4.00 (7.55) | 0.00 (1.29)
  Test 2: Baseline to Post Neutral Cue | -0.33 (3.28) | 0.17 (0.17)
  Test 4: Baseline to Post Drug Cue | -1.50 (0.50) | 0.33 (0.21)
  Test 4: Baseline to Post Neutral Cue | -7.00 (8.00) | -0.67 (0.67)

7. Secondary Outcome: Vital Signs - Heart Rate
Description: Heart rate (in beats/min) will be monitored throughout the time course of the study and changes from baseline will be studied across the various time points.
  **For test visits I, II and IV, there will be two cue sessions at each test visit: a neutral cue video (PN) and a drug-related cue video (PC) will be shown in random order at each visit. Before the beginning of each cue session (PN or PC), baseline measures will be taken. Heart rate will be measured again following the neutral cue video and the drug-related cue video. Thus there will be two sets of baselines and two sets of post cue measurements per test visit for test visits I, II and IV.
Time Frame: Test sessions 1,2,and 4: baseline 1, post cue (PC), baseline 2, post neutral cue (PN)
Measure: Mean (Standard Error); unit: beats per minute
Arm/Group | Control | CBD Group
Number analyzed (Participants) | 3 | 6
beats per minute
  Heart rate change (bpm): test 1 baseline to PC | -2.33 (1.67) | 4.00 (2.21)
  Heart rate change (bpm): test 1 baseline to PN | -6 (7.55) | 2.5 (2.72)
  Heart rate change (bpm): test 2 baseline to PC | -8 (3.06) | -6.5 (3.15)
  Heart rate change (bpm): test 2 baseline to PN | -1.33 (0.67) | -3.33 (2.5)
  Heart rate change (bpm): test 4 baseline to PC | 0 (1.15) | -3.33 (1.78)
  Heart rate change (bpm): test 4 baseline to PN | -1.67 (2.67) | -2.17 (2.5)

8. Secondary Outcome: Vital Signs - Respiratory Rate
Description: Respiratory rate (in breaths/min) will be monitored throughout the time course of the study and changes from baseline will be studied across the various time points.
  **For test visits I, II and IV, there will be two cue sessions at each test visit: a neutral cue video (PN) and a drug-related cue video (PC) will be shown in random order at each visit. Before the beginning of each cue session (PN or PC), baseline measures will be taken. Respiratory rate will be measured again following the neutral cue video and the drug-related cue video. Thus there will be two sets of baselines and two sets of post cue measurements per test visit for test visits I, II and IV.
Time Frame: Test sessions 1,2,and 4: baseline 1, post cue (PC), baseline 2, post neutral cue (PN)
Measure: Mean (Standard Error); unit: breaths per minute
Arm/Group | Control | CBD Group
Number analyzed (Participants) | 3 | 6
breaths per minute
  Respiratory rate (bpm): test 1 baseline to PC | 0 (0) | 0 (0.52)
  Respiratory rate (bpm): test 1 baseline to PN | 0 (0) | 0 (0.52)
  Respiratory rate (bpm): test 2 baseline to PC | -0.67 (0.67) | 0 (0.52)
  Respiratory rate (bpm): test 2 baseline to PN | 0 (0) | -1 (0.45)
  Respiratory rate (bpm): test 4 baseline to PC | -0.67 (0.67) | -0.67 (0.42)
  Respiratory rate (bpm): test 4 baseline to PN | -0.67 (0.67) | 0.33 (0.33)

9. Secondary Outcome: Vital Signs - Temperature
Description: Temperature (in degrees Fahrenheit) will be monitored throughout the time course of the study and changes from baseline will be studied across the various time points.
  **For test visits I, II and IV, there will be two cue sessions at each test visit: a neutral cue video (PN) and a drug-related cue video (PC) will be shown in random order at each visit. Before the beginning of each cue session (PN or PC), baseline measures will be taken. Temperature will be measured again following the neutral cue video and the drug-related cue video. Thus there will be two sets of baselines and two sets of post cue measurements per test visit for test visits I, II and IV.
Time Frame: Test sessions 1,2,and 4: baseline 1, post cue (PC), baseline 2, post neutral cue (PN)
Measure: Mean (Standard Error); unit: degrees F
Arm/Group | Control | CBD Group
Number analyzed (Participants) | 3 | 6
degrees F
  Temperature change (F): test 1 baseline to PC | 0.03 (0.03) | -3.35 (3.33)
  Temperature change (F): test 1 baseline to PN | 0.43 (0.75) | 0.03 (0.13)
  Temperature change (F): test 2 baseline to PC | 0.0 (0.1) | 0.05 (0.10)
  Temperature change (F): test 2 baseline to PN | 0 (0.2) | 0.02 (0.19)
  Temperature change (F): test 4 baseline to PC | 0.3 (0.31) | 0.18 (0.08)
  Temperature change (F): test 4 baseline to PN | 0.13 (0.28) | -0.17 (0.09)

ADVERSE EVENTS:
Description: Adverse events were collected by using SAFTEE (Systematic Assessment for Treatment Emergent Events)
Groups:
- CBD Group: Subjects received 400 mg or 800mg of cannabidiol.The two arms (400 mg and 800 mg CBD groups) were combined for analysis as CPD Group because the sample size was too small and dividing the two arms would not have yielded a meaningful analysis.
  Subjects in Arm CBD received 400 mg or 800mg of Cannabidiol in each of the three test sessions
Arm/Group | Control | CBD Group
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/6
Other Adverse Events (participants affected / at risk) | 3/3 | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=3) | CBD Group (N=6)
Diarrhea (Gastrointestinal disorders) | 1 (3) | 1 (1)
Dizziness (Vascular disorders) | 0 (0) | 1 (1)
Heavy Eyes (Nervous system disorders) | 1 (1) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 2 (2) | 0 (0)
Increased Appetite (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomach/abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1)
Increased Thirst (General disorders) | 1 (1) | 0 (0)
Drowsiness (Nervous system disorders) | 3 (3) | 1 (1)
Feeling down (Nervous system disorders) | 0 (0) | 1 (1)
Feeling irritable (Nervous system disorders) | 0 (0) | 1 (1)
Muscke/bone/joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Increased urine frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
Change in urine color (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less